CLINICAL TRIAL: NCT02835066
Title: A Pilot Study Investigating Patient Function/Fitness and Psychosocial Health in Patients With Non-Small Cell Lung Cancer
Brief Title: Patient Function/Fitness and Psychosocial Health in Improving Health-Related Quality of Life in Patients With Stage I-IV Non-Small Cell Lung Cancer
Status: Withdrawn | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CCCWFU 98515; NCI-2016-00649 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 98515 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2016-05-12; First posted 2016-07-15 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Smoking; Lung Neoplasms
Keywords: Stage I; Stage II; Stage IIIA; Stage IIIB; Stage IV; Non-Small Cell
MeSH Terms: conditions — Smoking; Lung Neoplasms | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (HRQOL, fitness and psychosocial health): Patients scheduled for surgery, radiation therapy, or chemotherapy complete the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-core 30 (C30) and QLQ-Lung Cancer 13 (LC13) in addition to psychosocial health and smoking status questions from baseline up to 2 weeks prior to the start of treatment, 5-6 weeks after treatment begins, and 5-6 months from the start of treatment. During the same time points, patients also undergo function/fitness assessments including standard health measurements, short physical performance battery (SPPB), 6 minute walk test (6MWT), and a grip strength test.
  Interventions: Other: Integrated Fitness Assessment; Procedure: Psychosocial Assessment and Care; Procedure: Quality-of-Life Assessment

INTERVENTIONS:
Other: Integrated Fitness Assessment — Undergo function/fitness assessment
Procedure: Psychosocial Assessment and Care — Undergo psychosocial health assessments
  Other Names: Psychosocial Assessment; Psychosocial Care; Psychosocial Care/Assessment; Psychosocial Studies; Psychosocial Support
Procedure: Quality-of-Life Assessment — Complete EORTC QLQ-C30 and QLQ-LC13 questionnaires
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot trial studies patient function/fitness and psychosocial health in improving health-related quality of life and decreasing treatment-related toxicity in patients with stage I-IV non-small cell lung cancer. Studying function/fitness and psychosocial health may help doctors improve conventional therapy in patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the correlation of patient-reported health-related quality of life (HRQOL) outcomes with clinical/treatment variables as well as a panel of both function/fitness and psychosocial health assessments in non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To investigate the panel of function/fitness and psychosocial health assessments with patient's smoking history/status as a predictor for treatment related toxicity.

TERTIARY OBJECTIVES:

I. The documentation of the NSCLC lung population from this prospective combined with others.

OUTLINE:

Patients scheduled for surgery, radiation therapy, or chemotherapy complete the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-core 30 (C30) and QLQ-Lung Cancer 13 (LC13) in addition to psychosocial health and smoking status questions from baseline up to 2 weeks prior to the start of treatment, 5-6 weeks after treatment begins, and 5-6 months from the start of treatment. During the same time points, patients also undergo function/fitness assessments including standard health measurements, short physical performance battery (SPPB), 6 minute walk test (6MWT), and a grip strength test.

After completion of study treatment, patients are followed up every 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed lung cancer

Exclusion Criteria:

* Previous or active lung cancer treatment at the time of registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Non-Small Cell Lung Cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Patient function/fitness | Up to 6 months
  Assessed by standard health measurements.
Patient well-being | Up to 6 months
  Assessed by questionnaires.
Patient function/fitness | Up to 6 months
  Assessed by performance-based measures.
Patient well-being | Up to 6 months
  Assessed by psychosocial health questions.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lally, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States